CLINICAL TRIAL: NCT02132169
Title: A Multi-Center, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety of AC-170 0.24% Ophthalmic Solution Used Twice Daily in Healthy Adult Subjects and in Pediatric Subjects With a History or Family History of Atopic Disease (Including Allergic Conjunctivitis)
Brief Title: A Multi-Center Study Evaluating the Safety of AC-170 0.24%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aciex Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-100-0006
Record Dates: First submitted 2014-04-29; First posted 2014-05-07 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Atopic Disease (Including Allergic Conjunctivitis)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AC-170 0.24% (Experimental)
  Interventions: Drug: Drug: AC-170 0.24%
- AC-170 0% (Placebo Comparator)
  Interventions: Drug: AC-170 0%

INTERVENTIONS:
Drug: Drug: AC-170 0.24%
  Other Names: 1 drop in each eye 2 times daily for up to 6 weeks
  Arms: AC-170 0.24%
Drug: AC-170 0%
  Other Names: 1 drop in each eye 2 times daily for up to 6 weeks
  Arms: AC-170 0%

SUMMARY:
The purpose of this study is to evaluate the safety of AC-170 0.24% used twice daily in Healthy Adult Subjects and in Pediatric subjects with a history or family history of atopic disease (including allergic conjunctivitis).

ELIGIBILITY:
Inclusion Criteria:

* at least 2 years of age
* be able to self-administer eye drops or have a parent/legal guardian available for this purpose
* if less than 18 years old have a history or family history of atopic disease (including allergic conjunctivitis)
* have ocular health within normal limits

Exclusion Criteria:

* known contraindications or sensitivities to the study medication or its components
* any ocular condition that, in the opinion of the investigator, could affect the subjects safety trial parameters
* use of disallowed medication during the period indicated prior to the enrollment or during the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey L Ackerman, MD, Principal Investigator — Philadelphia Eye Associates; Dawn K De Castro, MD, Principal Investigator — Andover Eye Associates; Edward J Meier, MD, Principal Investigator — Apex Eye; Eugene E Protzko, MD, Principal Investigator — Seidenberg Protzko Eye Associates
Locations (1):
- Ora, Inc., Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from four sites in the US.
Pre-assignment Details: There were 512 subjects enrolled, 24 subjects discontinued, and 488 subjects completed the study. Participant flow and baseline characteristics are presented for the 512 subjects that met all inclusion criteria and none of the exclusion criteria and were randomized to receive AC-170 0.24% or AC-170 0%.
Groups:
- AC-170 0.24%: 1 drop in each eye 2 times daily for up to 6 weeks AC-170 0.24%
- AC-170 0%: 1 drop in each eye 2 times daily for up to 6 weeks AC-170 0%
Period: Overall Study
Arm/Group | AC-170 0.24% | AC-170 0%
Started | 341 | 171
Completed | 326 | 162
Not Completed | 15 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AC-170 0.24% | AC-170 0% | Total
Number analyzed (Participants) | 341 | 171 | 512
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (19.36) | 36.6 (19.56) | 35.4 (19.42)
Age, Customized [Number; unit: participants]
  2-6 years old | 20 | 13 | 33
  7-12 years old | 28 | 12 | 40
  13-17 years old | 34 | 16 | 50
  >/= 18 years old | 259 | 130 | 389
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 114 | 309
  Male | 146 | 57 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 11 | 31
  Not Hispanic or Latino | 321 | 160 | 481
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 14 | 37
  White | 298 | 149 | 447
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 4 | 18
Region of Enrollment [Number; unit: participants]
  United States | 341 | 171 | 512

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of AC 170 0.24% Compared to Its Vehicle at Visit 1 (Day 1)
Description: Tolerability was assessed upon instillation of study medication, at 30 seconds and 1 minute post study medication instillation. Drop comfort was assessed using a 0-to 10 scale where 0=very comfortable and 10=very uncomfortable.
Time Frame: Upon instillation, 30 Seconds Post-Instillation, 1 minute Post-Instillation
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 341 | 171
units on a scale
  Upon instillation | 0.9 (1.36) | 0.5 (1.02)
  30 seconds post-instillation | 0.7 (1.25) | 0.3 (0.82)
  1 minute post-instillation | 0.6 (1.22) | 0.3 (0.75)

2. Primary Outcome: Tolerability of AC 170 0.24% Compared to Its Vehicle at Visit 2 (Day 8)
Description: as for outcome 1
Time Frame: Upon instillation, 30 Seconds Post-Instillation, 1 minute Post-Instillation
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 341 | 171
units on a scale
  Upon instillation | 0.8 (1.24) | 0.3 (0.80)
  30 seconds post-instillation | 0.5 (1.02) | 0.3 (0.74)
  1 minute post-instillation | 0.4 (0.90) | 0.2 (0.63)

3. Primary Outcome: Tolerability of AC 170 0.24% Compared to Its Vehicle at Visit 3 (Day 22)
Description: as for outcome 1
Time Frame: Upon instillation, 30 Seconds Post-Instillation, 1 minute Post-Instillation
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 341 | 171
units on a scale
  Upon instillation | 0.6 (1.13) | 0.2 (0.66)
  30 seconds post-instillation | 0.4 (0.83) | 0.2 (0.51)
  1 minute post-instillation | 0.3 (0.80) | 0.1 (0.47)

4. Secondary Outcome: Safety of AC 170 0.024% Compared to Its Vehicle
Description: Safety measures (adverse events) of AC 170 0.024% compared to its vehicle were measured at Visit 1-4 and 5 (for subset of patients).
Time Frame: Up to 12 Weeks
Population: Intent to Treat (ITT)
Measure: Number; unit: adverse events
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 341 | 171
adverse events | 70 | 40

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. All subjects who received study medication were evaluable for the safety analysis.
Description: Throughout the visits, staff collected all Adverse Events reported, elicited or observed.
Arm/Group | AC-170 0.24% | AC-170 0%
Serious Adverse Events (participants affected / at risk) | 1/341 | 1/171
Other Adverse Events (participants affected / at risk) | 65/341 | 39/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC-170 0.24% (N=341) | AC-170 0% (N=171)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC-170 0.24% (N=341) | AC-170 0% (N=171)
Conjunctival Hyperaemia (Eye disorders) | 27 (29) | 19 (20)
Ocular Hyperaemia (Eye disorders) | 10 (11) | 3 (3)
Vision Blurred (Eye disorders) | 2 (2) | 3 (3)
Dry eye (Eye disorders) | 1 (1) | 3 (3)
Visual acuity reduced (Eye disorders) | 2 (2) | 2 (2)
Eye discharge (Eye disorders) | 1 (1) | 2 (2)
Instillation Site Pain (General disorders) | 20 (21) | 3 (3)
Headache (Nervous system disorders) | 2 (3) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes